CLINICAL TRIAL: NCT02910076
Title: The Influence of Plaquenil/Hydroxychloroquine (HCQ) on Insulin Secretion
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0059-16-HMO-CTIL
Record Dates: First submitted 2016-09-01; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Type Two
MeSH Terms: interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy volunteers (Experimental)
  Interventions: Drug: Hydroxychloroquine
- Diabetes patients (Experimental)
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — 200 MG Plaquenil three times a day
  Other Names: Plaquenil

SUMMARY:
Antimalarials such as hydroxychloroquine (HCQ), are among the oldest prescribed drugs still used in clinical practice. Relatively inexpensive and well tolerated, these drugs have been recognized to be effective in autoimmune diseases such as rheumatoid arthritis (RA) and systemic lupus erythematosus (SLE). Interestingly, there is growing evidence of their beneficial impact on cardiovascular risk, particularly diabetes. HCQ therapy can improve balance in patients with unbalanced diabetes. This drug therapy may be a new therapeutic approach for diabetes. There is need for a better understanding of the mechanisms responsible for the improvement of the metabolic response to drug treatment. The investigators hypothesize that treatment with a drug improves the function of the beta cell and its ability to secrete insulin in response to glucose. The investigators will examine the impact of short-term therapy for HCQ in beta cell function in healthy volunteers and in patients with type 2 diabetes.

ELIGIBILITY:
Two groups will participate in this study: Healthy volunteers and Diabetes patients

A. Healthy volunteers

* Inclusion Criteria:

  * Age: 18-40
  * Without acute disease at the day of the experiment.
  * Signed informed consent
* Exclusion Criteria:

  * Malignancy
  * Steroids or NSAID on a daily basis

B. Diabetes patients

* Inclusion Criteria:

  * Age: 20-60
  * Diabetes type two
  * Untreated or on metformin treatment
* Exclusion Criteria:

  * Hypoglycemic medications

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
glucose level | the change in glucose level between baseline and after three hours